CLINICAL TRIAL: NCT02148432
Title: Establishment of Ideal IV Sedative Regimen for Successful Fiberoptic Bronchoscopy in Assessing the Site, Severity of Sleep Apnea Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 4-2014-0232
Record Dates: First submitted 2014-05-22; First posted 2014-05-28 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Sleep Apnea Syndrome
Keywords: sleep apnea syndrome, fiberoptic bronchoscopy, IV sedation
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexmedetomidine 0.5 mcg/kg/hr (Experimental)
  Interventions: Drug: dexmedetomidine infusion rate, 0.5 mcg/kg/hr
- dexmedetomidine 1.0 mcg/kg/hr (Active Comparator)
  Interventions: Drug: dexmedetomidine infusion rate, 1.0 mcg/kg/hr

INTERVENTIONS:
Drug: dexmedetomidine infusion rate, 0.5 mcg/kg/hr — continuous infusion of dexmedetomidine at rate of 0.5 mcg/kg/hr
  Arms: dexmedetomidine 0.5 mcg/kg/hr
Drug: dexmedetomidine infusion rate, 1.0 mcg/kg/hr — continuous infusion of dexmedetomidine at rate of 1.0 mcg/kg/hr
  Arms: dexmedetomidine 1.0 mcg/kg/hr

SUMMARY:
Venous thromboembolism(VTE) is the third most common cardiovascular complication among hospitalized patients, and can even cause death. VTE often occurs in intensive care patients and there had been many efforts to prevent such complication. The American College of Chest Physicians (ACCP) had published evidence-based clinical practice guideline for VTE prophylaxis.

This study focuses on how VTE prophylaxis is being performed in both medical and surgical ICUs in a single University hospital, and sees the differences in such prophylactic patterns.

ELIGIBILITY:
Inclusion Criteria:

1. 20-60 years old patients with ASA class I-II
2. Scheduled for drug induced sleep endoscope after diagnosed with sleep apnea syndrome

Exclusion Criteria:

1. Patients having hearing difficulties, taking any CNS related medication, history of any adverse drug reaction, Glasgow coma scale < 15
2. Patients with severe cardiopulmonary dysfunction
3. Patients refusal

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2014-05-19 (Actual); Primary Completion 2016-04-29 (Actual); Study Completion 2016-04-29 (Actual)

PRIMARY OUTCOMES:
Desaturation rate | Baseline from 5 min after remifentanil TCI start, 10 min after dexmedetomidine loading start, every 5 min until surgeon can do endoscopy successfully, to immediately after endoscopy
  SpO2 < 90% (checked by pulse oximetry)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Severance Hospital, Yonsei University College of Medicine, Seoul, Seoul, South Korea